CLINICAL TRIAL: NCT06237660
Title: Development of Non-invasive Biomarkers to Direct Individualised Management of Preschool Wheeze
Brief Title: Longitudinal Preschool Wheeze Biomarker Study
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Action Medical Research (Other); Masonic Charitable Foundation (Unknown); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23IC8468; GN3005 (Other Grant/Funding Number: Action Medical Research)
Record Dates: First submitted 2023-11-29; First posted 2024-02-01 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Wheezing
Keywords: Preschool wheeze; Preschool asthma; Allergy; Infection; Steroids
MeSH Terms: conditions — Respiratory Sounds; Hypersensitivity; Infections | interventions — Bronchoscopy; Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Bronchoalveolar lavage
  2. Endobronchial biopsy
  3. Blood
  4. Oropharyngeal swab
  5. Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Aim 1: To test the proposed panel of simple bedside tests below, to see how accurately they corelate with lower airway infection or inflammation.
  The aim is correlate the results from the bronchoscopy with the panel of test proposed, and evaluate if these simple bedside tests can pick up the same level of infection or inflammation and obtain the same results, as the bronchoscopy, which is a much more invasive test, but the only method available at present to get this information.
  Interventions: Procedure: Bronchoscopy, with bronchoalveolar lavage and endobronchial biopsy; Diagnostic Test: Skin prick test; Diagnostic Test: Finger prick blood test; Diagnostic Test: Forced oscillation technique (FOT); Procedure: Sputum induction; Diagnostic Test: Oropharyngeal swab
- Aim 2: The aim is to test how acceptable these bedside tests are to parents and children, and if they reflect the child's symptoms, symptoms control and medication use.
  Interventions: Diagnostic Test: Skin prick test; Diagnostic Test: Finger prick blood test; Diagnostic Test: Forced oscillation technique (FOT); Procedure: Sputum induction; Diagnostic Test: Oropharyngeal swab
- Aim 3: Small proof-of-concept study. This is for a feasibility trial of using the proposed tests and deciding the treatment of their wheeze, based on the results of the tests. Children with evidence of allergen sensitisation +/- blood eosinophilia (>0.3x109/L) will be prescribed regular inhaled corticosteroids. Children who are non-atopic (non-atopic is defined as blood eosinophil of <0.3x109/L + no evidence of allergen sensitisation) with positive bacterial detection in sputum, will be prescribed four weeks of targeted antibiotics. Children who are non-atopic with no bacteria detected in sputum, will be prescribed only be prescribed short acting bronchodilators as required. All medications will be prescribed, as per the British National Formulary for Children, based on age and weight.
  The aims of this preliminary study are to understand whether parents will agree to be part of such an interventional trial. This will help the research team when designing a future larger clinical trial.
  Interventions: Diagnostic Test: Skin prick test; Diagnostic Test: Finger prick blood test; Diagnostic Test: Forced oscillation technique (FOT); Procedure: Sputum induction; Diagnostic Test: Oropharyngeal swab

INTERVENTIONS:
Procedure: Bronchoscopy, with bronchoalveolar lavage and endobronchial biopsy — These children who will be having a bronchoscopy (a long thin tube, with a camera at the end, which is put inside the lung to look at and collect samples) as part of their standard clinical management, determined by their own consultants or treating physicians. They will be having lung samples (washings from the lung and a tiny piece of tissue taken from the breathing tubes) taken as part of their usual medical management. The research team will ask for consent to use the leftover samples for the bronchoscopy, for the study
  Groups: Aim 1
Diagnostic Test: Skin prick test — To identify children with allergies. This test will not be done if the child has had allergy testing in the last 6 months
Diagnostic Test: Finger prick blood test — Finger prick testing will be used for blood samples, and it is the same technique used by children with diabetes, to test their blood sugar levels, and therefore is regularly used in this age group successfully. The research team will be obtain the results within minutes, using a point-of-care device. A few more drops of blood, from the same finger prick sample, will be taken to look at how one of the blood cells work, in more detail, in the laboratory. There is no additional finger prick required for this lab test, and the drops of blood will be collected at the same time, from the same prick, as the point of care test.
Diagnostic Test: Forced oscillation technique (FOT) — Breathing test will be performed using forced oscillation technique (FOT), to see how the child's lungs work and to detect airway inflammation. The test will be explained to the child and completed using our established protocols. This test will only require the child to breathe in and out normally, and therefore can be done in preschool aged children. The current test that is used to check lung function called spirometry cannot be used in preschool children, as it involves following complicated instructions. The aim is to assess how well this newer lung function test is tolerated, in children aged 1-5 years.
Procedure: Sputum induction — Sputum induction is a test of obtaining phlegm after inhalation of salt water mist (saline nebuliser) and this will allow the research team to look for any relationships between infection in the lungs and the accuracy of the less invasive, nose and throat swabs. The research team will obtain phlegm samples, with a quick suction after patients have inhaled the salty mist (saline nebuliser) which will help loosen up their phlegm. If the child can cough it up, they will be encouraged to do it.
Diagnostic Test: Oropharyngeal swab — Swabs from children's nose and throats (similar to swab tests that are done for Covid tests), that will be used to test for bacterial infection

SUMMARY:
Preschool children (aged 1-5 years) account for 75% of all UK childhood wheezing hospitalisations. This has not changed over 20 years, meaning current treatments are not working and a new approach is needed. Currently, all preschool wheezers are treated with inhaled steroids. However, only about 25% of patients, with allergies, respond well to inhaled steroids; for the other 75%, they are ineffective. This research group has found that some preschool wheezers may have other causes but there are no specific, non-invasive tests to match the right treatment to each child.

The goal of this observational study is to test various bedside tests for this purpose in preschool children with wheeze, to see if they are feasible, accurate and acceptable in this age group.

The research team would like to investigate the following aims:

Aim 1 - To test the proposed panel of simple bedside tests below, to see how accurately they corelate with lower airway infection or inflammation.

Aim 2 - To test the acceptability of these bedside tests are to parents and children, and if they reflect the child's symptoms, symptoms control and medication use.

Aim 3- A small proof-of -concept study, to test if these simple bedside tests, can be used to determine treatment for each individual child.

The panel of simple non-invasive tests that the research team are proposing are:

1. Skin prick tests to common allergies (house dust mite, cat, dog, grass, tree pollen, mixed moulds)
2. Finger prick blood test
3. Phlegm test for bacteria
4. Nose and throat swab for bacteria
5. Lung function test called forced oscillation technique (FOT)

DETAILED DESCRIPTION:
Research Question:

Can the research team identify simple bedside tests that can give quick, accurate results while being acceptable to parents and children, and can these tests be successfully used in clinical practice, to decide treatment for preschool wheeze?

Participants will be asked to do these simple tests- skin prick test, finger prick blood test, breathing test, throat swab, and a test to catch their phlegm. The researchers will use two tests to identify children who are likely to respond to inhaled steroids: skin tests for allergies and a finger prick blood test. To identify children with bacterial infections in their lungs, where antibiotics will be useful, the team will obtain a sample of sputum (phlegm) after a salty mist inhalation (saline nebuliser), and will test the accuracy of a throat swab that detects bacteria. The research team will also test how cells called neutrophils work in children without allergies or infection with the same finger prick blood test above. A breathing test called forced oscillation will be used to identify children who may respond to their reliever "blue" inhaler during wheezing attacks.

The research team will also recruit a small number of children, for a trial in which their treatment will be guided by their test result, to see if parents are willing to take part in such a study, before designing a larger trial. This study will be the first to show that new tests can identify different types of preschool wheezing and can be used to plan treatment based on individual children's needs. Researchers will compare to see if children who have their treatment based on the simple bedside tests do better than the children who are just given inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

Aim 1, 2 and 3:

* Children aged 1-5 years
* More than 2 hospitalisations for acute wheeze in the last year or
* At least 1 admission requiring high dependency unit or intravenous bronchodilator therapy in the last year.

Aim 1 only:

- children undergoing clinically indicated bronchoscopy, as determined by their existing medical team, as part of their standard management

Exclusion Criteria:

* Alternative respiratory diagnosis such as cystic fibrosis or bronchiectasis.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitment will be from the Royal Brompton Hospital, which is a tertiary referral centre for respiratory paediatrics, but also receives direct referrals from GPs in North West London. This target population includes children from all sociodemographic and ethnic backgrounds as referrals are received from across London and the Southeast region.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal study of skin prick tests as biomarkers of preschool wheeze | 3 years
  Specificity, sensitivity and longitudinal stability of skin prick tests to six common allergens (measured by size of wheal in response to skin prick, measured in mm) as a biomarker of allergen sensitisation.
Longitudinal study of finger-prick point of care test for eosinophil count as a biomarker of preschool wheeze | 3 years
  Specificity, sensitivity and longitudinal stability of a finger-prick point of care test for eosinophil count (measured as cells per cubic mm) as a biomarker of eosinophilic inflammation.
Longitudinal study of blood neutrophil phenotype as a biomarker of airway infection | 3 years
  Specificity, sensitivity and longitudinal stability of blood neutrophil phenotype (measured as mean fluorescence intensity for indicative phenotype markers) as a biomarker of airway infection.
Longitudinal study of blood neutrophil chemotaxis as a biomarker of wheezing phenotype | 3 years
  Specificity, sensitivity and longitudinal stability of blood neutrophil chemotaxis (measured in micrometers per minute) as a biomarker of wheezing phenotype.
Longitudinal study of oropharyngeal swab and induced sputum PCR as a biomarker of airway infection | 3 years
  Specificity, sensitivity and longitudinal stability of oropharyngeal swab and induced sputum PCR (measured by detectable presence or absence of DNA from Haemophilus influenzae, Streptococcus pneumoniae and Moraxella catarrhalis) as biomarkers of airway infection. Concordance between oropharyngeal swab and induced sputum PCR results from the same patient will also be assessed.
Longitudinal study of lung function test (FOT) as a biomarker of airway reversibility | 3 years
  Specificity, sensitivity and longitudinal stability of lung function test (forced oscillation technique or FOT), measured by lung reactance and lung resistance (Rrs: respiratory system resistance; Xrs: respiratory system reactance; AX: area of reactance), as biomarkers of airway reversibility in wheezing patients.

SECONDARY OUTCOMES:
Association between eosinophil counts and patient symptom control | 3 years
  Measurement of eosinophil counts (measured as cells per cubic mm) in relation to patient symptom control, using the Test for Respiratory and Asthma Control in Kids (TRACK), a caregiver-completed validated questionnaire for preschool-aged children (measured as mean symptom score). TRACK is a 5-item standardized questionnaire, with each item being scored from 0 to 20 points on a 5-point Likert-type scale. Total score ranging from 0 to 100. Higher scores indicate better respiratory and asthma control; a score of less than 80 points suggests that a child's breathing problems might not be controlled.
Patient acceptability of finger prick blood eosinophil count as a non-invasive biomarker in preschool wheeze | 3 years
  Determining the patient acceptability of finger prick blood eosinophil count as a non invasive biomarker test, using the Visual Analogue Scale (VAS) of pain intensity. The scale ranges from 0 to 10, with 0 being no pain or discomfort and 10 for worst pain possible. Higher scores indicate worse tolerability.
Patient acceptability of skin prick test as a non-invasive biomarker in preschool wheeze | 3 years
  Determining the patient acceptability of skin prick test as a non invasive biomarker test, using the Visual Analogue Scale (VAS) of pain intensity. The scale ranges from 0 to 10, with 0 being no pain or discomfort and 10 for worst pain possible. Higher scores indicate worse tolerability.
Patient acceptability of forced oscillation technique as a non-invasive biomarker to determine lung function and airway reversibility in preschool wheeze | 3 years
  Determining the patient acceptability of forced oscillation technique as a non invasive biomarker test, to determine lung function and airway reversibility in preschool children, using the Visual Analogue Scale (VAS) of pain intensity. The scale ranges from 0 to 10, with 0 being no pain or discomfort and 10 for worst pain possible. Higher scores indicate worse tolerability.
Patient acceptability of oropharyngeal swab and induced sputum PCR as a biomarker of airway infection in preschool wheeze | 3 years
  Determining the patient acceptability of oropharyngeal swab and induced sputum PCR as a biomarker of airway infection in preschool children, using the Visual Analogue Scale (VAS) of pain intensity. The scale ranges from 0 to 10, with 0 being no pain or discomfort and 10 for worst pain possible. Higher scores indicate worse tolerability.
Correlation between eosinophil counts and symptom burden of preschool wheeze to caregivers | 3 years
  Correlation between measurement of eosinophil counts (measured as cells per cubic mm) and assessment of symptom burden of preschool wheeze to caregivers using the validated Paediatric Asthma Caregivers Quality of Life Questionnaire (PACQLQ), measured by mean life quality score. This is a questionnaire that is self-administered by the caregiver, and assess symptom burden to caregivers, across two domains (activity limitations and emotional function). Each question is assessed using a 7-point Likert scales, with 1 indicating severe impairment and 7 indicating no impairment. Domains scores are calculated as the mean score across items in that domain. The overall score is the mean score across all items. The lowest score achievable is 1 and highest score achievable is 7, and higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Saglani, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Clinical data that is needed for analysis and integration into the project will only be used in a pseudonymised fashion. All subjects will be given study identifier numbers. This data set as well as data dictionaries, will the be made available to the other members of the research team, eg, statisticians for data analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: Data sharing during the project will only be between researchers and collaborators involved in the project. Sharing with the wider scientific community will be enabled at the time of peer review and publication of the data. Secure and responsible data sharing will take place using file encryption and College, secure servers, requiring password protected access to the data.
  At the end of the project and after publication data will be made available for other researchers.
  Data sharing will be undertaken according to Imperial College guidance using a data sharing licence which will allow sharing data while stating clearly what others can do with the data.
  Tools such as License Selector that allow the best license for the type of data generated will be used to decide on the most appropriate licence for data and software.

REFERENCES:
- [Background] Robinson PFM, Fontanella S, Ananth S, Martin Alonso A, Cook J, Kaya-de Vries D, Polo Silveira L, Gregory L, Lloyd C, Fleming L, Bush A, Custovic A, Saglani S. Recurrent Severe Preschool Wheeze: From Prespecified Diagnostic Labels to Underlying Endotypes. Am J Respir Crit Care Med. 2021 Sep 1;204(5):523-535. doi: 10.1164/rccm.202009-3696OC. PMID 33961755

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT06237660/Prot_SAP_000.pdf